CLINICAL TRIAL: NCT06161051
Title: Treatment Patterns and Real-World Clinical Outcomes in Patients With Advanced NSCLC and MET Exon 14 Skipping Mutation in the United States
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CINC280AUS16
Record Dates: First submitted 2023-12-05; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Advanced Non-small Cell Lung Cancer and MET Exon 14 Skipping Mutation
Keywords: aNSCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- Capmatinib
- IO monotherapy
- Chemotherapy alone
- IO + chemotherapy

SUMMARY:
This was a retrospective, noninterventional cohort study of patients with a confirmed diagnosis of advanced non-small cell lung cancer (aNSCLC) with MET exon 14 skipping mutation who received treatment with capmatinib, immunotherapy (IO), or chemotherapy (CT) in real-world practice settings. Data abstraction was performed by the participating physician.

ELIGIBILITY:
Inclusion Criteria:

* Patient was aged ≥ 18 years at the time of NSCLC diagnosis.
* Had histologically confirmed advanced (stage IIIB, IIIC, or IV) NSCLC with MET exon 14 skipping mutation.
* Initiated first-line (1L) treatment for aNSCLC between 1 January 2017 and date of data abstraction with one of the following treatment regimen:

  * Capmatinib
  * IO agent in monotherapy (e.g., atezolizumab, pembrolizumab)
  * CT regimen, single agent or combinations of CT agents (e.g., platinum agents, taxane agents, gemcitabine, pemetrexed)
  * Combination regimen containing IO and CT agents
* Had ≥ 6 months of potential follow-up time after the initiation of 1L treatment for aNSCLC, except if the patient died sooner.
* Living or deceased at the time of chart abstraction.

Exclusion Criteria:

* Presence of other mutations (e.g., EGFR, ALK, ROS1, RET, NTRK, BRAF, or KRAS) at any time.
* Treatment with other MET inhibitors such as crizotinib or tepotinib at any time during the study period.
* Participation in clinical trials related to treatment for NSCLC at any timepoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Time-to-treatment discontinuation (TTD) | Up to approximately 5 years
Real-world overall response rate (rwORR) | Up to approximately 5 years
  Proportion of patients with best overall response of either a complete response (CR) or partial response (PR) to the line of therapy based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, or per healthcare professional (HCP) assessment.
Real-world disease control rate (rwDCR) | Up to approximately 5 years
  Proportion of patients with best overall response of either a CR+PR or stable disease to the line of therapy based on RECIST version 1.1, or per HCP assessment.
Real-world duration of response (rwDOR) | Up to approximately 5 years
  Time from the date of first documented CR or PR to the first documented systemic disease progression or death due to any cause.
Real-world progression-free survival (rwPFS) | Up to approximately 5 years
  Time from start of therapy until the earliest of a clinically documented systemic disease progression.
Overall survival (OS) | Up to approximately 5 years
  Time from start of therapy until death.

SECONDARY OUTCOMES:
Number of patients per demographic category | Baseline
  Demographic categories included sex, race/ethnicity, and insurance status.
Mean age | Baseline
Number of patients per clinical characteristic category | Baseline
  Clinical characteristics included staging, presence and site(s) of metastases, number of lesions, and performance status.
Number of patients per comorbidity | Up to 6 months pre-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States